CLINICAL TRIAL: NCT00626795
Title: Efficacy, Safety and Tolerability of TD1414 2% Cream in Impetigo and Secondarily Infected Traumatic Lesions (SITL)
Brief Title: Efficacy, Safety, and Tolerability of TD1414 2% Cream in Impetigo and Secondarily Infected Traumatic Lesions (SITL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TD1414-C21
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2018-08

CONDITIONS: Impetigo; Secondarily Infected Traumatic Lesions
MeSH Terms: conditions — Impetigo | interventions — Mupirocin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: TD1414 2% cream
- 2 (Experimental)
  Interventions: Drug: TD1414 2% cream
- 3 (Active Comparator)
  Interventions: Drug: Bactroban® (mupirocin) 2% cream

INTERVENTIONS:
Drug: TD1414 2% cream — BID 7 days
  Arms: 1
Drug: TD1414 2% cream — TID 7 days
  Arms: 2
Drug: Bactroban® (mupirocin) 2% cream — BID 7 days
  Arms: 3

SUMMARY:
An international, multi-centre, prospective three arm parallel-group, phase II proof of concept study comparing the efficacy and safety of two dosage regimens (BID 7 days and TID 7 days) of TD1414 2% cream and one dosage regimen (BID 7 days) of Bactroban® (mupirocin) 2% cream in adults and children down to 2 years of age with impetigo or SITL. Furthermore an evaluation of the pharmacokinetics of TD1414 2% cream TID for 7 days will be performed. A total of 664 patients will be enrolled in a stepwise manner according to age groups starting with the oldest age group.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent from patient and/or legally acceptable representative has been obtained
* Outpatients of any sex or ethnic origin
* Patients >= 2 years of age (depending on study step)
* Patients must be suffering from primary bullous/non-bullous impetigo or SITL

Exclusion Criteria:

* Presence of skin diseases at or near the investigational area
* Immunosuppressed state or other serious systemic disease
* Signs and/or symptoms of systemic infection
* Presence of skin infection/disorder not amenable to topical antibacterial treatment only
* Presence of secondarily-infected animal/human bite
* Presence of secondarily infected burnwound
* Topical or systemic use of medicinal or other products before or during the study which in the investigators opinion could confound the evaluation of the effect of the study drugs
* Known or suspected hypersensitivity to TD1414 or any of the excipients in the TD1414 2% cream
* Known or suspected hypersensitivity to mupirocin or any of the excipients in the Bactroban® (mupirocin) 2% cream
* Participation in any other investigational drug study or use of (an) investigational drug(s) within the 30 days or 5 half-lives (whichever is longer) prior to randomisation
* Patients previously enrolled/randomised in this study
* Abnormal ECG at baseline though the PR interval may be up to 220 ms, the QRS interval up to 110 ms and the QTc interval up to 450 ms

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 773 (Actual)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Almena L Free, MD, Principal Investigator — Anniston Medical Clinic
Locations (2):
- Anniston Medical Clinic, Anniston, Alabama, United States
- Division of Dermatology, Groote Schuur Hospital, G23, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An open-label treatment consisting of one arm with 4 age groups of 16 participants treated with TD1414 cream three times daily was used in a stepwise inclusion, to detect major safety issues that could prevent the study from proceeding. The participants in the open-label phase were not included the efficacy analysis or in the randomized population
Groups:
- TD1414 BID: TD1414 2% cream: two times daily (BID) 7 days
- TD1414 TID: TD1414 2% cream: three times daily (TID) 7 days
- Bactroban® TID: Bactroban® (mupirocin) 2% cream: three times daily (TID) 7 days
Period: Open-label TD1414 Cream TID Treatment
Arm/Group | TD1414 BID | TD1414 TID | Bactroban® TID
Started | 0 | 65 | 0
Completed | 0 | 64 | 0
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Blinded Treatment
Arm/Group | TD1414 BID | TD1414 TID | Bactroban® TID
Started | 204 | 205 | 205
Completed | 194 | 200 | 196
Not Completed | 10 | 5 | 9
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Unacceptable adverse event | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Other reasons | 2 | 0 | 2
Not completed — Missing reason for withdrawal | 5 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TD1414 BID | TD1414 TID | Bactroban® TID | Total
Number analyzed (Participants) | 204 | 205 | 205 | 614
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 65 participants were assigned to open-label TD1414 cream TID treatment for the purpose of safety evaluations.
  years
    Participants assigned to open-label TD1414 TID: number analyzed (Participants) | 0 | 65 | 0 | 65
    Participants assigned to open-label TD1414 TID |  | 18.4 (20.0) |  | 18.4 (20.0)
    Participants randomized to blinded treatment | 38.6 (14.8) | 36.3 (14.3) | 38.3 (15.3) | 37.7 (14.8)
Age, Customized [Count of Participants; unit: Participants] — Population: 65 participants were assigned to open-label TD1414 cream TID treatment for the purpose of safety evaluations.
  Participants
    Participants assigned to open-label TD1414 TID: number analyzed (Participants) | 0 | 65 | 0 | 65
    Participants assigned to open-label TD1414 TID: ≥16 years old | 0 | 17 | 0 | 17
    Participants assigned to open-label TD1414 TID: ≥12 to <16 years old | 0 | 16 | 0 | 16
    Participants assigned to open-label TD1414 TID: ≥6 to <12 years old | 0 | 16 | 0 | 16
    Participants assigned to open-label TD1414 TID: ≥2 to <6 years old | 0 | 16 | 0 | 16
    Participants randomized to blinded treatment: ≥16 years old | 193 | 194 | 195 | 582
    Participants randomized to blinded treatment: ≥12 to <16 years old | 11 | 11 | 10 | 32
    Participants randomized to blinded treatment: ≥6 to <12 years old | 0 | 0 | 0 | 0
    Participants randomized to blinded treatment: ≥2 to <6 years old | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 65 participants were assigned to open-label TD1414 cream TID treatment for the purpose of safety evaluations.
  Participants
    Participants assigned to open-label TD1414 TID: number analyzed (Participants) | 0 | 65 | 0 | 65
    Participants assigned to open-label TD1414 TID: Female |  | 35 |  | 35
    Participants assigned to open-label TD1414 TID: Male |  | 30 |  | 30
    Participants randomized to blinded treatment: Female | 97 | 93 | 110 | 300
    Participants randomized to blinded treatment: Male | 107 | 112 | 95 | 314
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 85 | 79 | 73 | 237
  South Africa | 119 | 126 | 132 | 377

OUTCOME MEASURES:

1. Primary Outcome: Participants With Clinical Cure According to Investigator's Assessment
Description: At end of treatment (Day 8), the participants had their impetigo/Secondarily Infected Traumatic Lesions (SITL) evaluated by the (sub)investigator.
  Investigator's assessment of severity of infections (SIRS).
  * Exudates/pus
  * Crusting
  * Erythema
  * Oedema
  * Tissue Warmth
  * Itching
  * Pain
  Each sign/symptoms of infection was assessed by use of the following 4-point scale:
  * 0 = absent
  * 2 = mild
  * 4 = moderate
  * 6 = severe
  The scores were summed up to a total SIRS score.
  Clinical cure was either of the following:
  * Total absence of signs and symptoms of impetigo/SITL OR
  * Improvement - total SIRS score reduced to <8 and all individual clinical signs/symptoms included in the SIRS score should have been ≤4.
  Clinical failure was either of the following:
  * Signs and symptoms of impetigo/SITL that did not meet the definition of clinical cure
  * Unable to determine (e.g. participants who refuse clinical examination or did not show at end of treatment or follow-up).
Time Frame: At end of treatment (Day 8)
Population: All participants randomized to blinded treatment who received at least one application of study medication were included in the efficacy analysis. Two participants (one from TD1414 BID and one from Bactroban® TID) did not receive any study medication and are therefore not included.
Measure: Count of Participants; unit: Participants
Groups:
- TD1414 BID: TD1414 2% cream: two times daily (BID) for 7 days
- TD1414 TID: TD1414 2% cream: three times daily (TID) for 7 days
- Bactroban® TID: Bactroban® (mupirocin) 2% cream: three times daily (TID) for 7 days
Arm/Group | TD1414 BID | TD1414 TID | Bactroban® TID
Number analyzed (Participants) | 203 | 205 | 204
Participants
  Clinical cure | 167 | 184 | 174
  Clinical failure | 36 | 21 | 30
Statistical Analysis 1: Comparison: TD1414 TID vs Bactroban® TID; Test type: Non-Inferiority — The lower confidence limit greater or equal to -12.5% indicates non-inferiority; Difference in percentage = 4.56, 95% CI 2-sided [-1.59 to 10.71] — Estimated using a Cochran-Mantel-Haenszel approach, stratifying by country and disease (impetigo/SITL)
Statistical Analysis 2: Comparison: TD1414 BID vs Bactroban® TID; Test type: Non-Inferiority — The lower confidence limit greater or equal to -12.5% indicates non-inferiority; Difference in percentage = -3.35, 95% CI 2-sided [-10.28 to 3.57] — Estimated using a Cochran-Mantel-Haenszel approach, stratifying by country and disease (impetigo/SITL)

2. Secondary Outcome: Participants With Clinical Cure According to Investigator's Assessment
Description: At follow up (Day 15), the participants had their impetigo/SITL evaluated by the (sub)investigator.
Time Frame: At follow up (Day 15)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TD1414 BID | TD1414 TID | Bactroban® TID
Number analyzed (Participants) | 203 | 205 | 204
Participants
  Clinical cure | 173 | 188 | 185
  Clinical failure | 30 | 17 | 19

3. Secondary Outcome: Participants With Clinical Cure According to Investigator's Assessment.
Description: At end of treatment (Day 8) and at follow-up (Day 15), the participants had their impetigo/SITL evaluated by the (sub)investigator.
Time Frame: At end of treatment (Day 8) and follow-up (Day 15)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TD1414 BID | TD1414 TID | Bactroban® TID
Number analyzed (Participants) | 203 | 205 | 204
Participants
  Clinical cure | 158 | 177 | 166
  Clinical failure | 45 | 28 | 38

4. Secondary Outcome: Participants With Bacteriological Cure According to Bacteriological Samples
Description: At baseline (Day 1), end of treatment (EOT), and follow-up (FU), the investigator obtained a bacteriological sample to base the assessment on.
  Bacteriological cure was either of the following:
  * Eradication of the baseline pathogen.
  * Presumed eradication of the baseline pathogen
  * Infection with a pathogen different from the baseline pathogen at EOT or FU and the participant was NOT symptomatic.
  Bacteriological failure was any of the following:
  * Documented lack of eradication of the baseline pathogen.
  * Documented relapse (re-infection) with the baseline pathogen
  * Documented super-infection, i.e. infection with a pathogen different from the baseline pathogen at EOT or FU, and the participants was symptomatic
  * Presumed persistence of baseline pathogen: Non-evaluable participants- participants who refused bacteriological examination or did not show at EOT or FU, and clinical failures who had no bacteriological sample to rule out bacterial infection.
Time Frame: At end of treatment (Day 8), follow-up (Day 15) and end of treatment and follow-up
Population: Only the randomized participants that were infected with S. aureus or S. pyogenes at baseline were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | TD1414 BID | TD1414 TID | Bactroban® TID
Number analyzed (Participants) | 110 | 121 | 118
Participants
  End of treatment (Day 8): Bacteriological cure | 66 | 80 | 94
  End of treatment (Day 8): Bacteriological failure | 44 | 41 | 24
  Follow-up (Day 15): Bacteriological cure | 74 | 85 | 102
  Follow-up (Day 15): Bacteriological failure | 36 | 36 | 16
  End of Treatment and follow-up: Bacteriological cure | 57 | 66 | 86
  End of Treatment and follow-up: Bacteriological failure | 53 | 55 | 32

5. Secondary Outcome: Participants With Clinical and Bacteriological Cure According to Investigator's Assessment and Bacteriological Samples
Description: At end of treatment (Day 8) and at follow-up (Day 15) the participants had their impetigo/SITL evaluated by the (sub)investigator.
  At baseline (Day 1), end of treatment (Day 8) and at follow-up (Day 15) the investigator obtained a bacteriological sample on which an assessment of bacteriological cure was based.
Time Frame: At end of treatment (Day 8), follow-up (Day 15) and end of treatment and follow-up
Population: All participants randomized to blinded treatment who received at least one application of study medication and were infected with S. aureus or S. pyogenes at baseline were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | TD1414 BID | TD1414 TID | Bactroban® TID
Number analyzed (Participants) | 110 | 121 | 118
Participants
  End of treatment (Day 8): Clinical and bacteriological cure | 59 | 76 | 88
  End of treatment (Day 8): Clinical or bacteriological failure | 51 | 45 | 30
  Follow-up (Day 15): Clinical and bacteriological cure | 70 | 79 | 99
  Follow-up (Day 15): Clinical or bacteriological failure | 40 | 42 | 19
  End of Treatment and follow-up: Clinical and bacteriological cure | 52 | 60 | 80
  End of Treatment and follow-up: Clinical or bacteriological failure | 58 | 61 | 38

6. Secondary Outcome: Participants With Clinical Cure According to Investigator's Assessment
Description: At Day 4 the participants had their impetigo/SITL evaluated by the (sub)investigator.
Time Frame: At Day 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TD1414 BID | TD1414 TID | Bactroban® TID
Number analyzed (Participants) | 203 | 205 | 204
Participants
  Clinical cure | 108 | 130 | 120
  Clinical failure | 95 | 75 | 84

ADVERSE EVENTS:
Time Frame: From Day 4 to Follow-up (Day 15) and Additional Follow-up (Day 14 after follow-up)
Description: All patients assigned to open-label treatment who received at least one application of the study medication (TD1414) and for whom the presence or confirmed absence of adverse events was available were included in the open-label analysis set. All participants randomized to blinded treatment who received at least one application of study medication and for whom the presence or confirmed absence of adverse events was available were included in the safety analysis set and analyzed for safety.
Groups:
- TD1414 TID >=16 Years; TD1414 TID >=12 to <16 Years; TD1414 TID >=6 to <12 Years; TD1414 TID >=2 to <6 Years: Open-label phase TD1414 2% cream: three times daily (TID) for 7 days
- TD1414 BID: Blinded treatment TD1414 2% cream: two times daily (BID) for 7 days
- TD1414 TID: Blinded treatment TD1414 2% cream: three times daily (TID) for 7 days
- Bactroban® TID: Blinded treatment Bactroban® (mupirocin) 2% cream: three times daily (TID) for 7 days
Arm/Group | TD1414 TID >=16 Years | TD1414 TID >=12 to <16 Years | TD1414 TID >=6 to <12 Years | TD1414 TID >=2 to <6 Years | TD1414 BID | TD1414 TID | Bactroban® TID
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/16 | 0/16 | 2/203 | 2/205 | 0/204
Other Adverse Events (participants affected / at risk) | 6/17 | 5/16 | 2/16 | 3/16 | 61/203 | 49/205 | 34/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TD1414 TID >=16 Years (N=17) | TD1414 TID >=12 to <16 Years (N=16) | TD1414 TID >=6 to <12 Years (N=16) | TD1414 TID >=2 to <6 Years (N=16) | TD1414 BID (N=203) | TD1414 TID (N=205) | Bactroban® TID (N=204)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Penetrating abdominal trauma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Shunt occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TD1414 TID >=16 Years (N=17) | TD1414 TID >=12 to <16 Years (N=16) | TD1414 TID >=6 to <12 Years (N=16) | TD1414 TID >=2 to <6 Years (N=16) | TD1414 BID (N=203) | TD1414 TID (N=205) | Bactroban® TID (N=204)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Aneamia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Long QT syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Application site irritation (General disorders) | 1 | 1 | 0 | 0 | 18 | 16 | 9
Application site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 5 | 1
Application site pruritus (General disorders) | 2 | 0 | 1 | 0 | 4 | 5 | 5
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Treatment failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Application site swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Condition aggravated (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 4 | 3 | 2
Impetigo (Infections and infestations) | 0 | 0 | 0 | 3 | 6 | 3 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 3 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 3 | 0 | 0
Tinea capitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Human bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 5
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 7 | 1 | 6
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ligament disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 2
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Company acknowledges the investigators' right to publish the entire results of the study, irrespective of outcome. The Company retains the right to have any publication submitted to the Company for review at least 30 days prior to the same paper being submit-ted for publication or presentation. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.